CLINICAL TRIAL: NCT03966521
Title: The British Society of Endovascular Therapy ConformabLe EndoVascular Aneurysm Repair (BSET-CLEVAR) Registry
Brief Title: The British Society of Endovascular Therapy ConformabLe EndoVascular Aneurysm Repair Registry
Acronym: BSET-CLEVAR
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: The British Society of Endovascular Therapy (BSET) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 19SM5135; IRAS Project ID: 260562 (Other: Health Research Authority)
Record Dates: First submitted 2019-05-22; First posted 2019-05-29 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Abdominal Aortic Aneurysm Without Rupture
Keywords: Endovascular aneurysm repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the BSET-CLEVAR Registry is to collect device-specific performance outcomes of the GORE® EXCLUDER® Conformable AAA Endoprosthesis with ACTIVE CONTROL System (EXCC device) in routine clinical treatment of patients with abdominal aortic aneurysm in the UK.

The novel EXCC device is an evolution of an established device allowing active shaping to conform to the specific patient aortic neck anatomy, with more accurate deployment, potentially greater neck coverage and better long term fixation/sealing. This may translate to improved effectiveness of this device over time, reducing the need for any further procedures. The primary aim of this study is to assess the degree of neck coverage by the EXCC device.

The British Society of Endovascular Therapy (BSET) has received funds from the stent manufacturer (W.L. Gore & Associates, Inc.) to conduct this study. BSET and the Sponsor (Imperial College London) have full responsibility for the design, conduct, analysis and reporting of the study.

DETAILED DESCRIPTION:
An abdominal aortic aneurysm (AAA) is a 'bulge' caused by weakness of the wall of the aorta (main blood vessel) in the section that travels down through the abdomen. An AAA can grow to a large size over time and it may burst (rupture), causing life-threatening internal bleeding. The standard method to prevent the AAA from bursting is to re-line the aorta with an artificial piece of rigid tubing called a stent that has been covered with material. This is inserted through the blood vessels from the artery in the groin to stop the aneurysm from expanding and restore normal diameter of the aorta. This is commonly known as a 'keyhole'or minimally invasive approach called endovascular aneurysm repair (EVAR).

There have been many advances in stent-graft technology to improve the accuracy and effectiveness of the EVAR procedure. A new design of an existing stent-graft that is currently being used in patients in many hospitals is the GORE® EXCLUDER® Conformable AAA Endoprosthesis with ACTIVE CONTROL (also known as EXCC Device). This new device allows the operator to shape the upper end of the device so that it may be placed into the aorta more accurately, conforming to the shape of the aorta, potentially improving the fixation and long-term sealing of the aneurysm, which may translate to a reduction in the need for further procedures.

This study is a prospective, multi-centre observational cohort registry of patients undergoing routine clinical treatment of AAA by the EXCC device. Recruitment will take place in 13 experienced UK centres with extensive EVAR experience. Up to 150 participants will be recruited in 30 months and followed-up to 1 year (participants will not undergo any procedure that is not part of their routine clinical care). Clinical data and device specific outcomes, including complications and re-interventions will be prospectively collected. In addition, the BSET-CLEVAR Registry Core Lab will evaluate both the pre-operative CT scan and the post-operative CT scan (obtained between 4 weeks and 3-months following EVAR), to assess the primary outcome of the study (endograft positioning accuracy and aortic neck coverage expressed as percentage of the total aortic neck assessed). Study outcomes will also include detailed analysis of pathological and anatomical features of the aneurysm and the EXCC device, which will be used for reporting the effectiveness of the graft. A detailed statistical analysis plan will be written prior to the final analysis.

The Study Co-ordinating Centre based at Imperial College London is responsible for the overall coordination of the Study, including monitoring of the overall study progress and review of study data accuracy (which, if necessary, may be checked by auditing the source data).

ELIGIBILITY:
Inclusion Criteria:

The patient is / has:

* Age 55 or more at the time of informed consent signature.
* Non-ruptured infra-renal AAA that requires treatment, and in the opinion of the Investigator, whose anatomy is adequate to receive or has already received the GORE® EXCLUDER® Conformable AAA Endoprosthesis with ACTIVE CONTROL System (EXCC device).
* A signed and dated Informed Consent Form signed by the patient either before or within 30 days of EXCC device implantation

Exclusion Criteria:

The patient is / has:

* Previous infra-renal aortic surgery
* Been treated in another aortic or thoracic medical device study within 1 year of study enrollment.
* Active infection
* Penetrating aortic ulcer or dissection or intramural haematoma in the treated segment
* Any clinically significant medical condition, which in the opinion of the investigator, may interfere with the study results or reduce life expectancy to <2 years
* In the opinion of the investigator unable or unwilling to comply with the requirements of the study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with abdominal aortic aneurysm who are suitable for endovascular repair of their AAA and are either being considered for or have received treatment by endoprosthesis implantation as part of their routine care at a participating NHS hospital
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Endograft positioning accuracy and aortic neck coverage expressed as percentage of the total aortic neck assessed by CT images | between 4 weeks and 3 months following EVAR
  The median aortic neck surface area utilized will be calculated from pre- and post-operative CT images, which will be obtained between 4 weeks and 3 months following primary EVAR procedure (timing depends on local EVAR surveillance policy)

SECONDARY OUTCOMES:
Technical success defined as successful access and deployment of all required EXCC Device components | At the end of the primary procedure
  (Yes/No) - Success defined as no type I/III endoleak, no conversion to open repair & patient leaving theatre alive; to be assessed by the operating clinician on completion of EVAR
In-hospital mortality | During hospital admission for the primary EVAR procedure, to be reported for up to 12 months following the primary procedure
  Death occurring during hospital stay for EVAR
Adjunct (supplementary) procedures received by the patient to resolve Type 1 endoleak on completion of EVAR | At the end of the primary EVAR procedure
  Further steps (procedures) required to deal with type 1 endoleak (a failure of the first section of the stent-graft as it is fixed in the aorta below the renal arteries)
Freedom from Type 1 or 3 endoleak | At the end of the primary procedure; at first follow-up (between 4 weeks and 3 months); at second follow-up (1 year)
  No type 1 endoleak (a failure of the first section of the stent-graft as it is fixed in the aorta below the renal arteries) or Type 3 endoleak (a failure of sealing of the components of the stent-graft)
One-year aneurysm-related re-intervention rate | One year after the primary procedure
  Any further aneurysm-related procedures that occur within 12 months following EVAR
One-year aneurysm-related mortality | One year after the primary procedure
  Vital status of the patient one year after undergoing EVAR

CONTACTS AND LOCATIONS:
Overall Officials: Colin D Bicknell, MB MD FRCS, Principal Investigator — Imperial College London
Locations (13):
- United Kingdom (13):
  - Hull & East Yorkshire Hospitals NHS Trust (Hull Royal Infirmary), Hull, East Yorkshire
  - Frimley Health NHS Foundation Trust, Frimley, Surrey
  - Imperial College Healthcare NHS Trust (St Mary's Hospital), London, Westminster
  - NHS Grampian, Aberdeen
  - Bedford Hospital NHS Trust, Bedford
  - University Hospitals Dorset NHS Foundation Trust, Bournemouth
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Gloucestershire Hospitals NHS Foundation Trust, Cheltenham
  - NHS Tayside, Dundee
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich

IPD SHARING:
Plan to Share IPD: Undecided